CLINICAL TRIAL: NCT03691428
Title: A Daily Self-Regulation Intervention for Persons With Early Stage Alzheimer's Disease and Related Dementias and Their Spouses
Brief Title: Stress Reduction Study for Partners of Early Stage Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000021852; R21AG055861-01A1 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-10-01 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Dementia Caregiving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Wish Outcome Obstacle Plan
- Wait-list (Other): Participants will get the WOOP training after the last outcome assessment.
  Interventions: Behavioral: Wish Outcome Obstacle Plan

INTERVENTIONS:
Behavioral: Wish Outcome Obstacle Plan — 1. Wish or goal: A wish (e.g. "responding calmly when the partner asks a question repeatedly"). 2. Outcome: The most positive outcome of realizing the wish or goal (e.g. "both partners feel respected and happy"). Then the participant vividly imagines the outcome. 3. Obstacle: The most critical internal, controllable, obstacle (e.g., "feeling impatient"). Then the participant vividly imagines the internal obstacle occurring. 4. Plan: The participant answers the following question: What action can I take or what thought can I think to overcome the obstacle (e.g., "take a deep breath, take my partner's perspective, and answer the question calmly"); then he or she forms an "if" [specified obstacle - when I feel impatient], "then I will" [specified action or thought to overcome obstacle - take a deep breath, take my partner's perspective, and answer the question calmly] plan.

SUMMARY:
This is a study designed to pilot a WOOP (Wish Outcome Obstacle Plan) intervention for spouses of persons with early stage dementia for the purposes of future research. The investigators will be using two cohorts. One who will get the intervention and the other who will be wait listed and receive the intervention at a later date. Spouses of persons with dementia will use WOOP, a brief goal attainment sequence, every day for 16 days. Participants will complete surveys before the intervention, at Day 16, and at a 3-month follow-up. The outcome measures are goal attainment, emotion regulation skills, psychological health, and support quality. As of 9/2020 this entire study is being conducted remotely.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* The couple is married or in a cohabiting, committed relationship.
* One partner has early Adult Dementia (AD) or a related dementia using criteria: symptoms consistent with early-stage dementia or memory impairment (e.g., AD, vascular dementia) and scores on the Neuropsychiatric Inventory (NPI) ≥3; Mini-Mental State Examination (MMSE) ≥18 and ≤27; and Barthel Index (BI) ≥5 and ≤1923. Or>20 on Telephone Interview for Cognitive Status. (TICS)
* The spouse will have to score 27 or higher on the MMSE. Or>25 on TICS.
* Both participants must agree to participate and complete baseline interviews.
* Both partners are at least 60 years old.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Joan Monin, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monin JK, Oettingen G, Laws H, David D, DeMatteo L, Marottoli R. A Controlled Pilot Study of the Wish Outcome Obstacle Plan Strategy for Spouses of Persons With Early-Stage Dementia. J Gerontol B Psychol Sci Soc Sci. 2022 Mar 3;77(3):513-524. doi: 10.1093/geronb/gbab115. PMID 34171086

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Wait-list
Started | 48 | 42
Completed | 42 | 34
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait-list | Total
Number analyzed (Participants) | 48 | 42 | 90
Age, Continuous [Mean (Full Range); unit: years] — Population: Ages of care partners and persons with dementia are presented individually.
  years
    care partners: number analyzed (Participants) | 24 | 21 | 45
    care partners | 72.3 [57 to 89] | 76 [60 to 89] | 74.0 [57 to 88]
    persons with dementia: number analyzed (Participants) | 24 | 21 | 45
    persons with dementia | 75.8 [60 to 99] | 77.2 [60 to 92] | 76.4 [63 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 23 | 20 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 43 | 39 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 48 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress
Description: The Perceived Stress Scale (PSS-10) will be used to examine participants' stress over the past week. There are 10 items rated on a scale from 0 to 4. Greater scores indicate greater stress. Sum scores can range from 0 to 40 with 40 being the highest stress and 0 being the lowest.
Time Frame: baseline, 3 months
Population: 3 month follow-up data for perceived stress was only provided by 21 care partners in the intervention condition and 17 in the wait-list condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait-list
Number analyzed (Participants) | 21 | 17
score on a scale | 13.6 (6.3) | 17.8 (13.6)
Statistical Analysis 1: Comparison: Intervention vs Wait-list; Test type: Superiority; p < .05, Mixed Models Analysis

2. Primary Outcome: Change in Positive Affect
Description: Nine self-reported positive emotions (e.g., amusement, gratitude, hope) on a 1-5 scale over the past week using the Positive and Negative Affect Schedule (25 items). Higher scores indicate more positive emotions. Mean scores can range from 1 to 5 with 5 being the highest experience of positive emotions.
Time Frame: baseline, 3 months
Population: 21 care partners in the intervention and 17 in the wait-list had positive emotion data at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait-list
Number analyzed (Participants) | 21 | 17
score on a scale | 3.60 (.61) | 3.20 (.87)
Statistical Analysis 1: Comparison: Intervention vs Wait-list; Test type: Superiority — A multivariate dyadic linear growth curve model was used to predict the trajectories of psychological well-being (Raudenbush, Brennan, & Barnett, 1995); p < .05, Mixed Models Analysis

3. Primary Outcome: Change in Depressive Symptoms
Description: 10-item Center for Epidemiologic Studies of Depression Scale (CESD). Participants rate on a scale from 0 to 3. Higher numbers indicate more depressive symptoms. Sum scores can range from 0 to 30 with higher sums cores meaning more depressive symptoms.
Time Frame: baseline, 3 months
Population: 20 caregivers in the intervention and 16 in the waitlist provided depression data at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-list
Number analyzed (Participants) | 20 | 16
units on a scale | 5.4 (5.07) | 9.75 (6.45)
Statistical Analysis 1: Comparison: Intervention vs Wait-list; Test type: Superiority; p < .05, Mixed Models Analysis

4. Primary Outcome: Change in Quality of Life
Description: Quality of life was measured with the Quality of Life in Alzheimer's Disease (QOL-AD). The QOL-AD consists of 13 items that capture multiple aspects of a person's quality of life in the context of dementia. It can also be used to examine the quality of life of family members of persons with dementia. Participants rate on a 5-point scale from poor to excellent the degree to which they feel about different aspects of their life (e.g. physical health, energy, mood, memory, family). Sum scores can range from 13 to 65 with higher scores meaning higher quality of life.
Time Frame: baseline, 3 months
Population: 21 care partners in the intervention and 17 in the waitlist group reported quality of life at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait-list
Number analyzed (Participants) | 21 | 17
score on a scale | 41.5 (6.9) | 35.5 (7.0)
Statistical Analysis 1: Comparison: Intervention vs Wait-list; Test type: Superiority; p < .05, Mixed Models Analysis

5. Primary Outcome: Change in Negative Emotions
Description: Ten negative (e.g., irritable, distressed) adjectives were measured with the Positive and Negative Affect Scale. Each item has a score of 1 (not at all) to 5 (extremely). The mean of the 10 items will be measured. Mean scores can range from 1 to 5 with 5 meaning the highest experience of negative emotions.
Time Frame: baseline, 3 months
Population: 21 care partners in the intervention and 17 in the waitlist reported negative emotions at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait-list
Number analyzed (Participants) | 21 | 17
score on a scale | 1.8 (.54) | 2.0 (.50)
Statistical Analysis 1: Comparison: Intervention vs Wait-list; Test type: Superiority; p < .05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention | Wait-list
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 0/48 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03691428/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03691428/SAP_001.pdf
  • Informed Consent Form (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03691428/ICF_002.pdf